CLINICAL TRIAL: NCT05344612
Title: Clinical Outcomes and Cost-effectiveness of a Diagnostic and Treatment Strategy of Upfront CTCA Plus Selective Non-invasive Functional Imaging Compared With Standard Care in Patients With Chest Pain and Suspected Coronary Artery Disease
Brief Title: Comparing a Diagnostic and Treatment Strategy of Upfront CTCA With SOC in Patients With Chest Pain and Suspected CAD
Acronym: CLEAR-CAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.P.S Henriques, Prof.Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL81264.018.22
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Chest Pain; CAD
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTCA (Experimental)
  Interventions: Radiation: CT Coronary Angiography
- Standard care (No Intervention)

INTERVENTIONS:
Radiation: CT Coronary Angiography — Upfront ct-coronary angiography
  Arms: CTCA

SUMMARY:
Rationale:

Patients with chest pain usually undergo multiple diagnostic examinations to demonstrate or rule out atherosclerotic coronary artery disease (CAD). In addition to high healthcare costs, some of the examinations do not assess the presence of CAD, which means that patients may be undertreated and are at risk for myocardial infarction. A uniform diagnostic and treatment strategy that uses computed tomography coronary angiography (CTCA) as initial examination may reduce major adverse cardiac events (MACE) and may reduce healthcare costs. In addition, we hypothesize that this strategy improves angina-related health status and reduces the number of invasive coronary angiograms (CAG's).

Objectives:

* To show that the intervention is non-inferior to the control with regards to clinical outcomes
* To show superiority of the intervention with regards to clinical outcomes

Study design: National multicenter prospective randomized controlled trial.

Study population: Patients with suspected stable CAD.

Intervention: upfront CTCA to diagnose CAD and guide optimal medical therapy (OMT). Patients with obstructive CAD and refractory angina despite OMT will undergo non-invasive ischemia imaging to guide revascularization.

Control: Standard of care. Diagnosis and treatment are at the discretion of the attending cardiologist.

Main study end point: Composite of all-cause mortality and non-fatal myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* >18 years

Exclusion Criteria:

* Presentation with acute coronary syndrome
* Acute coronary syndrome within last 3 months
* History of obstructive coronary artery disease on imaging
* History of PCI and/or CABG
* Severe renal failure
* Severe allergy to ionidated contrast medium
* Known pregnancy
* Patients with an estimated life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6444 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality and non-fatal myocardial infarction | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands